CLINICAL TRIAL: NCT00209144
Title: Effects of Intense Glycemic Control on Markers of Inflammation and Thrombosis in Patients Treated With Percutaneous Coronary Intervention for Acute Myocardial Infarction.
Brief Title: Phase 1 Study of Potential Anti-Inflammatory Effects of Glucose Control During Acute Myocardial Infarction.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Douglas Morris, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 867-2004; 6-56553
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Acute Myocardial Infarction
Keywords: Inflammation; Thrombosis; Hyperglycemia; Myocardial Infarction; Angioplasty
MeSH Terms: conditions — Inflammation; Thrombosis; Hyperglycemia; Myocardial Infarction

ARMS (2):
- Angioplasty with Insulin (Experimental): Coming in with acute infarct and received angioplasty with intensive insulin therapy
  Interventions: Drug: Intensive insulin therapy
- Angioplasty w/o Insulin (No Intervention): Coming in with acute infarct and received angioplasty

INTERVENTIONS:
Drug: Intensive insulin therapy
  Arms: Angioplasty with Insulin

SUMMARY:
The purpose of this study is to determine if intense control of high glucose levels in patients treated with angioplasty for heart attack has anti-inflammatory and anti-thrombotic effects.

DETAILED DESCRIPTION:
Two out of three heart attack patients have high blood sugar. Half of these patients have diabetes and the other half have what is called pre-diabetes, meaning that they have higher blood sugar than normal but not high enough to have diabetes. Over 40 million Americans have pre-diabetes.

For more than 70 years, doctors have known that patients with high blood sugar do not survive or recover from heart attacks as well as patients with normal blood sugar. Doctors have not figured out the reason for this difference.

The best treatment available for heart attacks is called angioplasty. Angioplasty means that doctors put a small balloon into a blocked blood vessel, blow up the balloon to open the blockage, and then insert a small wire tube called a stent to hold the blockage open. Blood thinners and other heart medicines are also given to these patients to help blood get through the blocked blood vessel. Angioplasty and these medicines have helped many people survive and recover from heart attacks. But even when doctors use these drugs, balloons and stents, patients who have high blood sugar still do worse than patients with normal blood sugar.

We want to figure out why high blood sugar is bad for patients with heart attacks. Past research tells us there might be two reasons. The first is that high blood sugar increases inflammation which is part of the body's natural response to heart attack. Inflammation is what causes a person's skin to turn hot and red after it is injured. Although inflammation is part of the body's natural healing process, too much inflammation can be harmful. We think that patients with high blood sugar during heart attacks have too much inflammation. The second reason why high blood sugar might be bad for heart attack patients is that high blood sugar makes blood thicker. When a blood vessel is blocked, thick blood makes it harder for the heart to get the blood flow it needs. This is why doctors use aspirin and other blood thinners when they treat patients with heart attacks.

The amount of inflammation and thickness in a person's blood can be measured in a laboratory. In this study, we want to measure the amount of inflammation and thickness in patients' blood to see if there is a difference between patients with normal blood sugar, patients with pre-diabetes, and patients with diabetes. If we can show that there is a difference, this will help us to understand why high blood sugar is bad for patients with heart attacks.

We also want to see if lowering a patient's high blood sugar is helpful during a heart attack. The standard therapy for lowering blood sugar in diabetic patients with heart attacks is to check their blood sugar four times each day while they are in the hospital, and to give them a shot of a medicine called insulin that helps bring the blood sugar level down if it is high. However, research tells us that this way of treating diabetic patients doesn't get their blood sugar low enough. Also, patients with pre-diabetes and patients who have diabetes but don't know it usually don't get any insulin, so their sugar levels are usually allowed to run high while they are in the hospital. In this study, we will treat half of diabetic and pre-diabetic patients the usual way and give the other half insulin through an IV for the first 24 hours that they are in the hospital. If we compare the inflammation and blood thickness between patients treated the usual way and patients treated with more insulin, we can figure out if lowering blood sugar more than usual is helpful to patients with heart attack.

If we can find out why high blood sugar is harmful to patients with heart attacks, and if we can show that treating these patients with more insulin than usual lessens these harmful effects, then we will be able to improve the way that these patients are treated. This could result in better survival and recovery for many heart attack patients.

All patients who volunteer for this study will get the best treatment available for heart attack- angioplasty, blood thinners, and the other heart medications that are usually given to these patients. Patients who have high blood sugar will be divided into two groups. One group will have their blood sugars measured and treated in the usual way. The other group will be treated with insulin run through an IV for 24 hours. After 24 hours, all patients will be treated in the usual way.

About one tablespoon of blood will be drawn from each patient at the time they sign up for the study and then 6, 12, 24, and 48 hours later. This blood will be used to test for inflammation and blood thickness.

The only ways in which patients who volunteer for this study will be treated differently from the standard of care are that they might receive more insulin than usual and they will have more blood drawn than usual. Giving extra insulin to these patients should not cause them harm, and may even help them. Since only about 5 tablespoons of extra blood will be drawn from each patient, this should not cause patients any harm.

Goals of this study

1. To see what happens to blood inflammation and thickness in heart attack patients with normal blood sugar and compare this to patients with high blood sugar.
2. To find out lowering patients' blood sugar levels more than we currently do will result in less blood inflammation and thickness.

ELIGIBILITY:
Inclusion Criteria: Patients to be treated with percutaneous coronary intervention for myocardial infarction.

Exclusion Criteria: MI > 6 hrs duration Thrombolytic therapy (within last 2 days) Recent inflammatory/infectious illness (last 2 weeks) Pregnancy Renal insufficiency (Cr > 2.0) Type I Diabetes Mellitus Initial BG >110 but <140 Enrollment in another research study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2004-10; Primary Completion 2005-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Troponin levels | Baseline, 24 hours, 48 hours, and 72 hours (post-procedure)

SECONDARY OUTCOMES:
CRP level | Baseline, 24 hours, 48 hours, and 72 hours (post-procedure)
B-type natriuretic peptide levels. | Baseline, 24 hours, 48 hours, and 72 hours (post-procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas C Morris, MD, Principal Investigator — Emory Heart Center
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - Emory Crawford Long Hospital, Atlanta, Georgia